CLINICAL TRIAL: NCT03904940
Title: Effectiveness of Total Contact Insole in Chronic Nonspecific Low Back Pain: a Randomized Controlled Trial
Brief Title: Total Contact Insole for Chronic Nonspecific Low Back Pain (LBP)
Acronym: (LBP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Anamaria Jones, Head of Rheumatology Rehabilitation Section - Rheumatology Division, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Federal University Sao Paulo
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: Orthotic Devices; Insoles; Quality of life; Function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total Contact Insole Group (Experimental): Ethyl vinyl acetate insole shaped in the cast of the patient's foot, every 6 months.
  Interventions: Device: Total Contact Insole
- Flat Insole group (Sham Comparator): Flat insole made the same material ethyl vinyl acetate, every 6 months.
  Interventions: Device: Ethyl vinyl acetate flat insole

INTERVENTIONS:
Device: Total Contact Insole — Ethyl vinyl acetate insole shaped in the cast of the patient's foot.
  Other Names: Intervention foot orthoses group
  Arms: Total Contact Insole Group
Device: Ethyl vinyl acetate flat insole — Flat insole made of the same material ethyl vinyl acetate
  Other Names: Placebo insole; Ethyl vinyl acetate flat insole group
  Arms: Flat Insole group

SUMMARY:
Non-specific low back pain is a common condition. Insoles are one of the many treatment form for chronic nonspecific LBP. The investigators hypothesized the contact total insole group will present pain reduction and functional improvement.

The aim of this study is to assess the effectiveness of contact total insole for people with nonspecific chronic low back pain and the impact of this insole on function, quality of life, load distribution in the plantar region, gait variables and satisfaction with insole use.

DETAILED DESCRIPTION:
A randomized, controlled, double-blind, clinical trial with intent-to-treat analysis. Eighty-four patients with nonspecific chronic low back pain will be randomly into a study group and control group. One week following the baseline evaluation, the study group will receive a contact total insole made of ethyl vinyl acetate and the control group will receive a flat insole made of the same material, color and density. The groups will be evaluated after 6, 12 and 24 weeks of insole use. The following assessment parameters will be employed: low back pain numerical pain scale; functional capacity (Oswestry and roland morris questionnaire, six minute walk test and timed to up and go test); quality of life (Short Form-36) and foot pressure analysis using the AMCube FootWalk Pro program.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain for more than 3 months, with numeric pain scale between 3 - 8 cm;
* Over 18 years;
* No distinction of sex;
* Understand Portuguese well enough to be able to fill in the questionnaires;
* Agree to participate of the study and sign the informed consent form.

Exclusion Criteria:

* Inflammatory/rheumatological diseases, tumor, infection or vertebral fracture;
* Litigation;
* Fibromyalgia;
* Other symptomatic musculoskeletal diseases in lower limbs;
* Symptomatic diseases of the central and peripheral nervous system;
* Diabetes Mellitus;
* Rigid deformities on foot;
* Use of insoles in the last three months;
* Medical or physiotherapeutic treatment for low back pain or any problem in lower limbs in the last three months;
* People who had changed physical activity or undergone physical therapy in the previous 3 months;
* Pregnancy;
* Difference of lower limbs greater than 2 cm
* Less than 6 months after lumbar spine, lower limb or abdomen surgery
* Previous spinal surgery;
* Previous spinal infiltration for pain relief in the last 3 months;
* Serious scoliosis;
* Allergy to the material of the insole.
* Planned travel in the next 12 weeks;
* Geographic inaccessibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Low back of pain intensity measured with Numeric Pain Rating Scale | Baseline, 45, 90 and 180 days
  It will be measured by the Brazilian version of the Numeric Pain Rating Scale 10 cm. The Numeric Pain Rating Scale goes from 0 to 10, where 0 is "no pain" and 10 is "the worst pain imaginable." Participants will be asked to answer about their pain levels based on the last week. Change in pain score or an improvement of 2 levels or more is accepted as clinically relevant.

SECONDARY OUTCOMES:
Functional capacity measured with Oswestry Disability Index | Baseline, 45, 90 and 180 days
  Change in Oswestry Disability Index score. Ranging from 0 to 100 with higher values represent a worse outcome
Functional capacity measured with Roland Morris Disability | Baseline, 45, 90 and 180 days
  Change in Roland Morris Disability score. Ranging from 0 to 24 with higher values represent a worse outcome
Functional capacity measured with the 6-minute walk test | Baseline, 45, 90 and 180 days
  Change in 6-minute walk test. The amount of meters walked in 6 minutes.
Functional capacity measured with the timed to up and go test | Baseline, 45, 90 and 180 days
  Change in timed to up and go test. Amount of time that the patient takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Quality of life measured with Short form-36 questionnaire | Baseline, 45, 90 and 180 days
  Change in Short form-36 questionnaire score. Ranging from 0 to 100 with higher scores showing a better outcome.
Patient's global impression of recovery measured with a likert scale | 45, 90 and 180 days after baseline
  The Likert scale. The patients answered the question 'After starting the use the insoles, how do you think your low back is?' with one of the following statements: much worse, a little worse, unchanged, a little better, much better.
Amount Medication consumption | 45, 90 and 180 days after baseline
  Amount of paracetamol (500mg) consumed by patient between the evaluation times
Foot pressure analysis using the AMCube FootWalk Pro program | baseline, 90 and 180 days after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil